CLINICAL TRIAL: NCT00816634
Title: A Randomized Phase II Trial of Capecitabine Plus Cisplatin (XP) Versus Capecitabine Plus Paclitaxel (XT) as a First-line Treatment for Advanced or Recurrent Esophageal Squamous Cell Carcinoma
Brief Title: Efficacy Comparison Study of Combination Regimens to Treat Advanced Esophageal Squamous Cell Carcinoma
Acronym: XP versus XT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young-Hyuck Im, professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-07-059
Record Dates: First submitted 2008-12-30; First posted 2009-01-01 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: First Line Chemotherapy; Capecitabine Plus Cisplatin Versus Capecitabine Plus Paclitaxel; Advanced or Recurrent Esophageal Squamous Cell Carcinoma
Keywords: First line chemotherapy; Advanced or recurrent esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Capecitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Chemotherapy regimen (XP):
  D1- D14 Capecitabine 1000 mg/m2 bid p.o. D1 Cisplatin 75 mg/m2 + NS 150mL MIV over 1hr repeat every 3 weeks
  Interventions: Drug: Capecitabine plus cisplatin(XP) versus capecitabine plus paclitaxel(XT)
- 2 (Active Comparator): XT Regimen:
  D1- D14 Capecitabine 1000 mg/m2 bid p.o. D1, D8 Genexol (Paclitaxel) 80 mg/m2 + D5W 500mL MIV over 3hrs Repeat every 3 weeks
  Interventions: Drug: Capecitabine plus cisplatin(XP) versus capecitabine plus paclitaxel(XT)

INTERVENTIONS:
Drug: Capecitabine plus cisplatin(XP) versus capecitabine plus paclitaxel(XT) — 3.2 Overview of Study Design This study is a prospective, randomized, phase II study comparing response rate between patients with XP chemotherapy versus XG chemotherapy for patients with metastatic squamous cell carcinoma.
  Chemotherapy regimen (XP):
  D1- D14 Capecitabine 1000 mg/m2 bid p.o. D1 Cisplatin 75 mg/m2 + NS 150mL MIV over 1hr every 3 weeks
  Chemotherapy regimen (XT):
  D1- D14 Capecitabine 1000 mg/m2 bid p.o. D1, D8 Genexol (Paclitaxel) 80 mg/m2 + D5W 500mL MIV over 3hrs every 3 weeks

SUMMARY:
Until today, the 5-FU/cisplatin combination is the reference regimen with 30-45% response rates, which is most commonly used to treat patients with metastatic, recurrent or locally advanced, unresectable squamous cell carcinoma of the esophagus. Because the classical dose schedule of this two-drug combination is cisplatin 100 mg/m2 day 1 and 5-FU 1000 mg/m2/day continuous infusion for 96-120 hr, prolonged administration time and mucosal toxicity are inconvenient to the patients with the aim of palliation. Capecitabine, which is oral prodrug of 5-FU and mimic continuously-infused 5-FU, is being investigated in phase I, II and III trials for the treatment of gastric, gastroesophageal, and esophageal cancers, primarily in the first-line metastatic setting. In our experience, capecitabine plus cisplatin combination (XP) as a first-line treatment for 45 patients with advanced or recurrent esophageal squamous cell carcinoma demonstrated a promising anti-tumor activity with 57% of response rate and showed tolerable toxicity with convenience.

Paclitaxel has been also investigated as monotherapy and in combination with cisplatin in patients with advanced esophageal cancer. A Dutch phase II study demonstrated that paclitaxel combination with carboplatin had shown an encouraging confirmed response rate of 59% with 51 patients with resectable esophageal cancer in neoadjuvant setting. Another Dutch phase II study showed 43% of response rate including 4% of CR with 8 months of response duration when paclitaxel plus cisplatin administration was given for patients with metastatic esophageal cancer. Although recently first-line palliative chemotherapy regimen in esophageal cancer has been investigated, many trials have failed to show superiority to 5-FU/cisplatin combination. Since we considered that XP or XT is more effective and convenient chemotherapy regimen than 5-FU/cisplatin, this randomized phase II study was planned to compare XP with XT in terms of efficacy and tolerability.

DETAILED DESCRIPTION:
1. Introduction and Study Rationale

   1.1 Esophageal squamous cell carcinoma Esophageal cancer is the seventh most common cancer in Korea, with almost 400,000 new patients diagnosed annually worldwide. There are large variations in the predominant histological type throughout the world but the majority of worldwide esophageal cancers are squamous cell carcinoma arising from the upper and middle thirds of the esophagus. Esophageal cancer is a highly virulent disease with a five-year survival rate of 10-15% . Metastatic esophageal carcinoma is an incurable disease with median survival duration of 6 to 8 months .

   1.2 5-FU plus Cisplatin (FP) combination chemotherapy Cytotoxic chemotherapy has been used to control tumor growth, improve quality of life and prolong survival although a survival advantage for chemotherapy over best supportive care alone in patients with metastatic cancer of the esophagus has not been proven in randomized trials. Although there is no standard chemotherapy regimen for metastatic esophageal cancer, various kinds of chemotherapy regimens have been used to alleviate symptoms caused by cancer and prolong survival and improve quality of life. Various phase-II trials have been performed to evaluate the effect of such chemotherapy. The activity of conventional single agent chemotherapy has been studied for cisplatin, 5-FU and mitomycin, which induced response rates of 15-30% . In most of these studies, the chemotherapy regimen consisted of a combination of cisplatin with another agent such as 5-FU or etoposide for both squamous cell carcinoma and adenocarcinoma. The most commonly used chemotherapy regimen for patients with advanced esophageal cancer is a combination of 5-FU and cisplatin, with response rates ranging from 15% to 45%, however, the effect on survival remained undetermined.

   1.2 Capecitabine for esophageal cancer Capecitabine is a novel, orally administered fluoropyrimidine carbamate that is absorbed readily by the gastrointestinal tract and is metabolized by the liver, where it is converted initially to 5 -deoxy-5-fluorocytidine (5 -DFCR) and subsequently, to 5 -deoxy-5-fluorouridine (5 -DFUR). Designed to mimic continuous intravenous (CIV) 5-FU, oral capecitabine predominantly concentrates in tumor tissue . Capecitabine currently is approved as a single agent for the adjuvant treatment of stage III colon cancer, as first-line treatment for metastatic colorectal cancer, and for metastatic breast cancer both as a single agent for patients and in combination with docetaxel. Whether oral fluoropyrimidines may be appropriately substituted, therefore making the therapy less burdensome to the patient and reducing the need for infusion catheters, is not fully investigated In patients with advanced esophagogastric cancer, capecitabine combinations have generally shown good antitumor activity and highlight the potential of capecitabine as a replacement of infusional 5-FU . Capecitabine has been investigated in combination with cisplatin and docetaxel in phase II trials in patients with advanced esophageal cancer with observed response rates of 47.1% and 46%, respectively . In a recent phase III trial comparing the efficacy of capecitabine/cisplatin (XP) versus FP in advanced gastric cancer, XP was not inferior to FP, in terms of progression-free survival (PFS), overall survival (OS), and response rate (RR) . In our experience, the combination of capecitabine and cisplatin for esophageal cancer showed encouraging response rate (59%) with tolerable toxicities and convenience.

   1.3 Paclitaxel for esophageal cancer Paclitaxel in combination with cisplatin has shown favorable results for advanced esophageal carcinoma . A recent phase II study of bi-weekly administration of paclitaxel and cisplatin in 51 patients resulted in complete response in 4%, partial response in 39%, stable disease in 43% and progressive disease in 14% of patients, and a one-year survival of 43% . Several phase II trials have assessed combinations of taxanes (paclitaxel and docetaxel) and cisplatin and other agents, with response rates of 40-56% .

   1.4 Capecitabine plus Paclitaxel combination for esophageal cancer Capecitabine in combination with docetaxel has greater efficacy than single-agent docetaxel; the combination increased survival significantly compared with single-agent docetaxel (14.5 v 11.5 months) in patients with metastatic breast cancer who experienced disease progression after anthracycline therapy . The most common treatment-related adverse events (TRAEs), with capecitabine 1,250 mg/m2 bid and docetaxel 75 mg/m2 were alopecia, hand-foot skin reaction (HFS), nausea, and fatigue. Neutropenia (15%) and HFS (11%) were the only grade 3 or 4 TRAEs that occurred in more than 10% of patients. In this trial the tolerable delivered dose of capecitabine for most patients was 950 mg/m2 bid for 14 days. Lorenzen et al. treated 24 patients with capecitabine at a dose of 1000 mg/m2 twice daily on Days 1 through 14 and docetaxel 75 mg/m2 on Day 1 of 3-week cycles. The RR was 46% and median survival was 15.8 months. However, the toxicity profile was high with two 2 treatment-related deaths, a high incidence of Grade 3 or 4 neutropenia (42%), and a high incidence of Grade 3 HFS (29%).

   There is a theoretical advantage to using paclitaxel on a weekly schedule in conjunction with capecitabine based on the duration of the upregulation of thymidine phosphorylase (dThPase) by paclitaxel in model systems. The metabolism of capecitabine to the active agent, FU, provides insight into the rationale for combining capecitabine with taxanes in this phase II study . The rationale for combining paclitaxel with capecitabine is based on the upregulation of dTHPase, which has been demonstrated in a model of athymic mice bearing capecitabine-resistant human colon cancer xenografts. Treatment with paclitaxel led to a 7.9-fold increase in intratumoral dThPase. An increase in dThPase activity occurred 4 days after treatment with paclitaxel and persisted for 10 days . These data led to the current concept for this clinical trial, using paclitaxel on days 1 and 8 during a 14-day exposure to capecitabine in patients with MBC. Moreover, these agents have nonoverlapping toxicities and therefore can be combined with reasonable tolerability. It was anticipated that by allowing a week off from weekly paclitaxel therapy, the frequency of sensory neuropathy could be reduced.

   Given the high degree of efficacy of the docetaxel/capecitabine combination, but the significant toxicity observed with 1,250 mg/m2 bid capecitabine schedule, as well as the promising efficacy and safety observed with weekly paclitaxel/capecitabine in the phase I study by Uhlmann et al [27], we choose weekly paclitaxel for combination regimen with capecitabine. Practically, our study regimen is capecitabine plus paclitaxel(XT) combination chemotherapy.

   1.5 XP vs XT for esophageal cancer Based on the rationale and our experience, we are going to conduct randomized phase II trial for metastatic esophageal cancer to evaluate the efficacy and feasibility comparing XP with XT.
2. Study Objectives

2.1 Primary Objective: To evaluate response rate for each treatment group (XP vs XT) for metastatic esophageal cancer.

2.2 Secondary Objectives:

1. toxicity
2. progression-free survival
3. quality of life
4. overall survival
5. predictive marker study influencing response and survival

3. Study Design 3.1 Randomization

1. Timing of randomization: Randomization will be performed after inclusion of the patient
2. Stratification factor: performance status (ECOG 0, 1 vs 2) & weight loss of 10% or more

3.2 Overview of Study Design This study is a prospective, randomized, phase II study comparing response rate between patients with XP chemotherapy versus XT chemotherapy for patients with metastatic squamous cell carcinoma.

Chemotherapy regimen (XP):

D1- D14 Capecitabine 1000 mg/m2 bid p.o. D1 Cisplatin 75 mg/m2 + NS 150mL MIV over 1hr Pre & Post medication D0 N/S 1500 mL IV overnight hydration D1 DNK2 1000 mL IV over 2 hours, pre & post hydration (if Mg < WNL, mix MgSO4 1 amp) 5-HT3 antagonist 1 amp + dexamethasone 20 mg + D5W 100 mL MIV 20% Mannitol 70 mL IV full dripping, 30 mins before cisplatin D2-D5 5-HT3 antagonist 1T QD D2-D3 Dexamethasone 8 mg PO bid D4-D5 Dexamethasone 4 mg PO bid every 3 weeks

Chemotherapy regimen (XT):

D1- D14 Capecitabine 1000 mg/m2 bid p.o. D1, D8 Paclitaxel 80 mg/m2 + D5W 500mL MIV over 3hrs Pre & Post medication D1, D8 Solucortef 100 mg IV push before Paclitaxel Avil 1A + D5W 50mL MIV 30mins before Taxol Ranitidine 50mg IV + D5W 50mL MIV 30mins before Paclitaxel HT3 antagonist 1A + D5W 50 mL MIV 30mins before Paclitaxel Followed by 1 week off every 3 weeks

3.3 Study Duration and Dates The duration of this study is expected to be 36 months, with subject recruitment proposed to start in October 2008. The actual overall study duration or subject recruitment period may vary.

3.4 Number of Patients/Assignment to Treatment Groups 94 patients will be recruited in total. Patients will be randomized to a treatment arm by permutated method. Chemotherapy should be started within 14 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic, or recurrent esophageal squamous cell carcinoma
2. Age > 18 years
3. ECOG performance status 0 - 2
4. At least one measurable lesion(s) by RECIST criteria
5. Life expectancy ≥ 3 months
6. Patients may have received prior adjuvant chemotherapy with 5-FU with cisplatin as long as it has been 12 months since completion of regimen.
7. No previous palliative chemotherapy
8. Prior radiotherapy must be completed 4 weeks before study entry.
9. Adequate bone marrow function (≥ ANC 1,500/ul, ≥ platelet 100,000/ul, ≥ Hemoglobin 9.0 g/dl)
10. Adequate renal function (≤ serum creatinine 1.5 mg/dl or CCr ≥ 50 ml/min)
11. Adequate liver function (≤ serum bilirubin 1.5 mg/dl, ≤ AST/ALT x 3 upper normal limit)
12. Written informed consent

Exclusion Criteria:

1. Other tumor types such as adenocarcinoma, small cell carcinoma
2. Evidence of CNS metastasis
3. Contraindication to any drug contained in the chemotherapy regimen
4. Previous adjuvant treatment with 5-FU, cisplatin, capecitabine or paclitaxel finished less than 1 year
5. Evidence of serious gastrointestinal bleeding
6. History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
7. Clinically significant cardiac disease (e.g. severe non-compensated hypertension, non-compensated heart failure, dilated cardiomyopathy, and coronary heart disease with ST segment depression in ECG) or myocardial infarction within the last 6 months.
8. Serious pulmonary conditions/illness (e.g. chronic lung disease with hypoxemia)
9. Serious metabolic disease such as severe non-compensated diabetes mellitus
10. History of significant neurologic or psychiatric disorders
11. Serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease
12. Positive serology for the HIV
13. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2008-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Response rates of both regimens | December 2010

SECONDARY OUTCOMES:
a) progression-free survival b) quality of life c) toxicity d) overall survival e) predictive markers | December 2010

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea